CLINICAL TRIAL: NCT06534502
Title: A Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Zonisamide Oral Suspension (100 mg/5 ml) to Determine a Dosing Regimen in Children 1 Month to 17 Years of Age With Partial-onset Seizures
Brief Title: Study of the Pharmacokinetics, Safety, and Tolerability of ZONISADE in Children 1 Month to 17 Years of Age With Partial-onset Seizures
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Azurity Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZ04.001
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Seizures; Seizures, Focal; Seizure, Partial Onset; Seizure Disorder, Partial; Seizure, Partial; Epilepsies, Partial; Epilepsy
Keywords: Partial-onset (focal) seizures; Pediatrics; ZONISADE; Zonisamide
MeSH Terms: conditions — Seizures; Epilepsies, Partial; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zonisamide Oral Suspension (Experimental): Zonisamide Oral Suspension, 100 mg/5 ml administered orally twice daily
  * Titration Period: 1 mg/kg/day administered as a divided dose of 0.5 mg/kg twice daily for 2 weeks, then increased by 1 mg/kg/day (as divided doses) at weekly intervals in Weeks 3 to 8.
  * Maintenance Period: Up to 8 mg/kg/day given as a divided dose twice a day for 4 weeks (i.e., Weeks 9 to 12).
  Interventions: Drug: Zonisamide Oral Product

INTERVENTIONS:
Drug: Zonisamide Oral Product — Zonisamide oral suspension
  Other Names: ZONISADE; Zonisamide oral suspension

SUMMARY:
The purpose of this research is to determine the optimal dose, safety and tolerability of zonisamide oral suspension in children ages 1 month to 17 years of age who have partial-onset (focal) seizures. The study consists of four periods: a Screening Period (about 14 days), a Titration Period (8 weeks), a Maintenance Period (4 weeks), and a Follow-Up Period (1 week).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric participants (ages 1 month to 17 years of age, inclusive) will be considered eligible for the study based on the following criteria:

  1. Voluntarily obtained informed consent from parent/legal guardian of the participant and assent from the participant, when appropriate.
  2. Willing and able to follow protocol specific requirements.
  3. Participant of 1 month to 17 years of age, inclusive (at time of consent).
  4. Participant diagnosed with partial-onset (focal) seizures, with or without secondary generalization as per current International League Against Epilepsy (ILAE) classification of seizures. Participants with both focal-onset and generalized-onset seizures are eligible, but only focal-onset seizures count toward baseline seizure enrollment criteria. Tonic-clonic and tonic seizures with unknown onset are presumed to be focal-onset unless there are clear clinical and EEG data suggesting generalized-onset.
  5. Participant with seizure occurrence more than once in the past three (3) months and more than two (2) times in the past six (6) months.

     a. Participant who is 6 months of age and younger will have seizure profiling patterns assessed by the Investigator for appropriate consideration and inclusion in the study.
  6. Participant on a stable regimen of anti-epilepsy drugs (AEDs) for at least 30 days before screening

     a. Participant who is 6 months of age and younger will have regimen assessed for inclusion in the study at Investigator's discretion.
  7. Participant with acceptable laboratory investigations:

     1. Hemoglobin within normal range
     2. Alanine aminotransferase (ALT) within normal range
     3. Aspartate aminotransferase (AST) up to 1.5 x upper limit of normal (ULN)
     4. Bilirubin within normal range
     5. Creatinine clearance within normal range
  8. If male participant is able to father children must be willing to use a highly effective method of contraception for at least one month after the last dose of investigational product if at risk of pregnancy with her/his partner. If female participant has reached menarche, the participant is authorized to participate in this clinical study if additional criteria are met.

At screening:

1. (i) Participant reports sexual abstinence for the prior 3 months or reports use of at least 1 of the acceptable methods of contraception, including an intrauterine device, barrier methods (e.g., male or female condom), hormonal contraceptives (e.g., hormonal patches, vaginal devices, oral pills), levonorgestrel intrauterine system (e.g., Mirena®), or regular medroxyprogesterone injections (e.g., Depo-Provera®); or (ii) Participant agrees to initiate sexual abstinence from the time of screening until at least one month after end of treatment with study drug; and
2. Participant is advised to avoid conception from the time of screening until at least one month after last receipt of study drug and agrees not to attempt pregnancy from the time of screening until at least one month after end of treatment with study drug; and
3. Participant is provided guidelines regarding continuation of abstinence, initiation of abstinence, or about allowed contraception; and
4. Participant has a negative serum β-human chorionic gonadotropin (β-hCG) test just prior to study entry. Since serum tests may miss an early pregnancy, relevant menstrual history and sexual history, including methods of contraception, should be considered. Note: if the result of the serum β-hCG test cannot be obtained prior to dosing of investigational product, a participant may be enrolled on the basis of a negative urine pregnancy test, though a serum β-hCG test result must still be obtained.

Exclusion Criteria:

* Pediatric participant will be excluded from the study based on the following criteria:

  1. Known hypersensitivity to zonisamide or to any component of the investigational product or to sulfonamides.
  2. Participant who is pregnant or nursing.
  3. Participant with exclusively generalized-onset seizures.
  4. Participant with predisposition to nephrolithiasis or prior history of kidney stone(s).
  5. Participant who is underweight (weight-for-age <2 standard deviation (SD) from the median of the World Health Organization (WHO) Child Growth Standards) or have a decreased appetite.
  6. Participant currently on or scheduled to receive carbonic anhydrase inhibitors such as topiramate or acetazolamide.
  7. Participant currently on or are scheduled to receive drugs known to have pharmacokinetic (PK) interaction.
  8. Participant who has previously received zonisamide.
  9. Participant with positive serology for Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), or Human Immunodeficiency Virus (HIV).
  10. Participant who has degenerative or metabolic disease of the brain.
  11. Participant with history of psychiatric disorder (excluding stable attention deficit hyperactivity disorder (ADHD), mood disorder on adequate treatment).
  12. Participant has any condition which, in the Investigator's opinion, would make it unsafe for the participant to participate in this study.
  13. Participant who has participated in other clinical study 30 days prior to enrollment in this study or 4-5 half lives of investigational drug, whichever is longer.
  14. Participant who uses alcohol or is currently on or scheduled to receive other central nervous system (CNS) depressants.
  15. Participant has a positive COVID-19 polymerase chain reaction (PCR) test result; or has had exposure (within 2 weeks prior to screening) to someone who had a positive COVID-19 test result; or is suspected of having long COVID-19 by the Investigator or designee.
  16. Participant who is missing more than 15% of daily diary entries during the screening period.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Concentration of serum zonisamide | Up to 15 weeks
  The concentration in serum of zonisamide following administration of zonisamide oral suspension, 100 mg/5 ml

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Up to 15 weeks
  Incidence of treatment-emergent adverse events (TEAEs), serious and non-serious, reported throughout the study.
Number and/or percentage of participants who discontinued the study because of adverse events | Up to 15 weeks
  Number and/or percentage of participants who discontinued the study because of adverse events
Number and/or percentage of participants who required zonisamide dose reduction because of TEAEs. | Up to 15 weeks
  Number and/or percentage of participants who required zonisamide dose reduction because of TEAEs.

OTHER OUTCOMES:
Change from baseline in seizure frequency | Up to 15 weeks
  Change from baseline in seizure frequency

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Le Bonheur Children's Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No